CLINICAL TRIAL: NCT03578614
Title: Randomized Interventional Prospective Study of the Effect of Physical Activity in Vascular Cognitive Impairment
Brief Title: Impact of Physical Activity in Vascular Cognitive Impairment ( AFIVASC )
Acronym: AFIVASC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Instituto de Medicina Molecular João Lobo Antunes (Other)
Collaborators: Fundação para a Ciência e a Tecnologia (Other)
Responsible Party: Principal Investigator, Ana Verdelho, Principal Investigador, Clinical Professor, Neurologist, Instituto de Medicina Molecular João Lobo Antunes
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: FCT-PTDC/DTP-ES/3706/2014
Record Dates: First submitted 2018-05-24; First posted 2018-07-06 (Actual); Last update posted 2021-04-01 (Actual); Status verified 2021-03

CONDITIONS: Vascular Cognitive Impairment
Keywords: Vascular cognitive impairment; Physical Activity; Randomized Clinical Trial; Stroke; TIA; Small Vessel Disease
MeSH Terms: conditions — Motor Activity; Stroke | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: Single-blind, randomized controlled trial, with a six-month intervention treatment and an additional follow-up of six months. After a four-week run-in period, the participants are randomized into two parallel groups (control group and intervention group).
Who Masked: Investigator
Masking Description: Single-blind
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (No Intervention): There is no intervention for Control Group
- Intervention Group (Experimental): Intervention Group will be submitted to three physical activity sessions (two supervised and one nonsupervised) conducted over 6 months
  Interventions: Other: Physical Activity

INTERVENTIONS:
Other: Physical Activity — 3 physical activity sessions are planned by week, 2 supervised and 1 non-supervised conducted over 6 months. On the first 2 months, the supervised sessions have 10 minutes of warm-up + 5 minutes active pause (balance, agility and coordinative exercises) + 15 minutes walking + 5 minutes active pause (resistance exercises - 1 series of 12 repetitions
  - 3 callisthenic exercises) + 15 minutes walking + 5 minutes flexibility (1 series of 10 seconds in 3 different postures). The aimed intensity in these first two months is 12/13. Between the 2nd and the 4th months, the duration of the walking period increases, as well as the intensity, RPE 13/14. Between the 4th and the 6th months, again the duration of the walking period increases, as well as the intensity, RPE 14/15. To measure the intensity level of the physical activity, the Borg Rating of Perceived Exertion (RPE) ranging from 6 (rest) to 20 (maximum effort) is used.
  Arms: Intervention Group

SUMMARY:
Vascular cognitive impairment (VCI) is one of the most frequent causes of cognitive impairment associated with aging. So far, there is no approved treatment for VCI. Recent studies have suggested a protective effect from physical activity but adequate studies are lacking in this field. The AFIVASC study - a Portuguese acronym for "physical activity in vascular cognitive impairment" is a randomized controlled study, single-blinded, nonpharmacological which aims to explore the benefits of physical activity in vascular cognitive impairment (VCI)

DETAILED DESCRIPTION:
Vascular cognitive impairment is one of the most frequent causes of cognitive impairment associated with aging. Vascular cognitive impairment includes clinical deficits due to vascular subclinical brain injury, silent lesions or due to clinically overt stroke, and appears frequently associated with Alzheimer disease. Vascular cognitive impairment has a spectrum of manifestations, from mild to extreme manifestation (Vascular Dementia) that represents the second most frequent cause of dementia. There is no approved treatment for vascular cognitive impairment, and pharmacological trials have generated disappointing results. As a result, nowadays, treatment is solely based on the control of vascular risk factors.

Walking is a physical activity recommended for the prevention of coronary disease. Besides, it is a physical activity without additional costs, easily accessible to the general population, and can be used in the whole population. Physical activity can potentially prevent functional decline associated with aging and promote global health status. In recent years, a growing interest has been given to the impact of physical activity as a protective factor for cognitive decline and for the progression for dementia There are several explanations for the protective effect in cognition: physical activity can implicate a better physical and global mental status, but can also be mediated through metabolic, physiopathological effects, as the increase cerebral inflow, the reduction of vascular risk factors, the decrease of production of stress hormones or still better endothelial function, among others.

However, there is no consensus in this field.

Some studies showed a protective effect of physical activity in Alzheimer disease. Protective effect of physical activity on vascular cognitive impairment (including dementia) has still to be proved. There are small studies with short follow-up, that do not take in consideration relevant confounding factors or imaging data (e.g. evidence of small vessel disease) with controversial results.

Recently a large observational study showed the beneficial impact of physical activity (defined according to the American Heart Association as at least 30 minutes of physical activity at least 3 times a week) in the reduction of the risk of progression for vascular dementia, in a cohort of subjects older than 65 years old, living independently, with cerebral white matter changes, and controlling for confounding factors. Additionally, in subjects with evidence of small vessel disease and no cognitive decline, physical activity was associated with better executive performance overtime.

The existing studies do not come from adequate randomized and double-blind designs, so there is no evidence-based data to sustain a recommendation for the type, intensity or frequency of physical activity, and the long-term gain. Given these contradictory findings, it becomes relevant to have an evidence-base to recommend physical activity in vascular cognitive impairment and in what concerns the type, intensity, and frequency of activity which would be necessary to achieve longterm gains.

ELIGIBILITY:
Inclusion Criteria:

* Participants are included if they are older than 18 years
* Fluent in Portuguese language;
* Able to read and write;
* Availability of a reliable informant;
* Fulfill the written informed consent;
* Clinical and functional criteria A and B:
* Criteria A: 1 of the following 3:

  1. Probable mild cognitive vascular impairment;
  2. Previous ischemic or hemorrhagic stroke (at least 6 months before), with modified Rankin ≤ 2 at baseline and without formal indication for physiotherapy.
  3. TIA (at least more than a 1 month before), diagnosed by a neurologist or with identified vascular lesion (correlated with TIA clinical symptoms) in CT/MRI.
* Criteria B: No functional changes: IADL 0 (no item changed, or 1 single item with minimal change), according to the scoring methods of the LADIS study (minimum of 4 items applicable) or no cognitive changes regarding the suggested Montreal Cognitive Assessment Test (Moca) cut off point for dementia in clinical Portuguese samples (score < 17).

Exclusion Criteria(Subjects cannot be included if they have at least one of the following):

* Diagnosis of dementia;
* Stroke with formal indication for physiotherapy or speech therapy, or Rankin ≥ 2;
* Any contraindication for walking, physical limitation to gait (orthopedic or other structural) that compromises the therapy proposed, or physical or mental limitation that could potentially interfere with the active treatment proposed (e.g. severe arthritis, severe osteoarticular pain associated with walking);
* Evidence of neurodegenerative disease (other than vascular aetiology), significant psychiatric disease (e.g. major depressive episode) or medical disease with prognosis or severity which could significantly interfere with the subjects' participation, or with quality of life (e.g. cancer, severe cardiovascular disease as congestive heart failure, uncontrolled angina).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 104 (Actual)
Dates: Start 2016-09-01 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2020-06-30 (Actual)

PRIMARY OUTCOMES:
Clinical Cognitive Criteria | 1 year
  Defined by a transition to dementia (all types) in patients with vascular cognitive impairment no dementia or transition to vascular cognitive impairment no dementia in those subjects with previous stroke/TIA without criteria for vascular cognitive impairment no dementia. This cognitive criteria will be assessed by a clinical neurologist
Cognitive Status measured by neuropsychological measures | 1 year
  Change in neuropsychological evaluation (1.5 SD of initial medium score) for composite scores calculated by averaging all different domains of the tests applied or for global measures (MOCA).

SECONDARY OUTCOMES:
Impact of physical activity in interpersonal, environmental, functional, physical, and psychological domains (Quality of Life) measured by Portuguese version of Quality of Live scale in Alzheimer's disease (QOL-AD) | 1 year
  Change in Quality of life (1.5 SD of initial medium score, using the Portuguese version of Quality of Life - Alzheimer Disease). The scale is composed of 13 items, quoted on a 4-point Likert scale, with higher scores indicating greater quality of life. The scale covers the domains: physical health, energy level, moods, living situation, memory, family, marriage, friends, overall self, ability to do chores around the house, ability to do things for fun, money, and overall life.
Impact of physical activity in motor status | 1 year
  Decline in activity performance (decrease in Fullerton Fitness Test, Fullerton Advanced Battery or reduction in gait velocity: 6 meters) according to the initial score.
Impact of physical activity in functional status | 1 year
  Decline in functional status (decrease in any item of the Instrumental Activities of Daily Living scale (IADL) - change from no change to any change or from minimal change to other change. Participants are scored according to their highest level of functioning in that category. A summary score ranges from 0 (low function, dependent) to 8 (high function, independent).

CONTACTS AND LOCATIONS:
Locations (1):
- Instituto de Medicina Molecular João Lobo Antunes, Lisbon, Portugal

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Verdelho A, Correia M, Ferro JM, Madureira S, Vilela P, Rodrigues M, Borges M, Oliveira V, Santos AC, Goncalves-Pereira M, Santa-Clara H. Physical Activity Self-Report Is Not Reliable Among Subjects with Mild Vascular Cognitive Impairment: The AFIVASC Study. J Alzheimers Dis. 2022;87(1):405-414. doi: 10.3233/JAD-215381. PMID 35275531
- [Derived] Verdelho A, Madureira S, Correia M, Ferro JM, Rodrigues M, Goncalves-Pereira M, Goncalves M, Santos AC, Vilela P, Barrios H, Borges M, Santa-Clara H. Impact of physical activity in vascular cognitive impairment (AFIVASC): study protocol for a randomised controlled trial. Trials. 2019 Feb 11;20(1):114. doi: 10.1186/s13063-019-3174-1. PMID 30744681